CLINICAL TRIAL: NCT00350883
Title: Cognitive Therapy for Negative Symptoms and Functioning
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Aaron T Beck, Universtiy of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 804915
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Cognitive Therapy; Negative Symptoms; Functional Outcomes; Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Behavioral Therapy; Therapeutics; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (Other)
  Interventions: Other: Treatment as Usual
- Cognitive Therapy (Experimental)
  Interventions: Behavioral: Cognitive Therapy

INTERVENTIONS:
Behavioral: Cognitive Therapy — Goal-oriented talk therapy
  Other Names: Cognitive Behavioral Therapy
  Arms: Cognitive Therapy
Other: Treatment as Usual — Keep getting usual care
  Other Names: Standard care; Enriched care
  Arms: Treatment as Usual

SUMMARY:
This clinical trial tests the effectiveness of cognitive therapy (CT) to improve outcomes in outpatients diagnosed with schizophrenia or schizoaffective disorder who manifest prominent negative symptoms. It is hypothesized that patients receiving cognitive therapy will manifest lower negative symptom levels and improved engagement in constructive activity relative to patients who receive treatment-as-usual. Further, it is predicted that these differences between CT and TAU will be larger when patients are assessed 6 and 12 months after the end of treatment (18 and 24 months after study entry).

DETAILED DESCRIPTION:
This is a clinical trial to evaluate the efficacy of adjunctive cognitive behavioral therapy for negative symptoms and functioning in chronic outpatients diagnosed with schizophrenia or schizoaffective disorder. After a baseline assessment to ensure eligibility, seventy-five consenting patients will be randomly assigned to receive a year of cognitive therapy (CT) or to a treatment as usual (TAU) control condition. Measures of symptomatology (positive, negative and affective), functioning, neurocognition and negativistic beliefs will be administered to all participants during five formal assessment sessions to occur at 6-month intervals over the course of a two-year period. The first assessment session (Baseline) will occur shortly after (i.e., within a week, though typically on the same day) informed consent is given. If the participant qualifies for the study and is consents to randomization, assessments identical to the baseline in content will occur 6, 12, 18 and 24 months later. All evaluators will be blind to participant treatment condition at the time of assessment.

The cognitive behavioral treatment will, in a collaborative and problem solving manner, target inaccurate or overly pessimistic expectations and thoughts about social and non-social performance. This psychosocial intervention will also target beliefs and attitudes that are related to positive symptoms which, in turn, exacerbate negative symptoms and impair functioning. We hypothesize that patients in the CT condition will have lower negative symptom levels and elevated functioning as compared to the TAU patients at the post-treatment assessment. Additionally, we expect that CT-treated patients will continue to improve over the follow-up period and, thereby, to continue to manifest lowered negative symptoms and elevated levels of functioning relative to TAU patients.

While research over the past 10 years has demonstrated the efficacy of CT as an adjunct intervention in the treatment of schizophrenia, negative symptoms have not been targeted directly, nor has an emphasis been placed upon improving functional outcomes. Given that negative symptoms and functioning are particularly refractory in this population, there is a need for treatment innovation. In this vein, our previous research (Grant & Beck, 2006) established that defeatist attitudes regarding social and non-social performance are important mediators in the causal chains that link neurocognitive performance, negative symptoms, and functional outcomes in schizophrenia. The current trial, thus, aims to move therapy for schizophrenia forward by improving long-term outcomes for some of the most impaired individuals in psychiatric service.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient diagnosed with schizophrenia or schizoaffective disorder
* Prominent negative symptoms (i.e., two global subscales rated "moderate" or higher on the Scale for the Assessment of Negative Symptoms
* Proficiency in English
* Able to give informed consent

Exclusion Criteria:

* Neurologic disease or damage
* Systematic medical illnesses that may compromise neurocognitive functioning (e.g., insulin dependent diabetes, heart disease)
* History of head injury or documented loss of consciousness
* Physical handicaps that would interfere with assessment procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Global Assessment Scale | baseline, 6 month, 12 month, 18 month, 24 month

SECONDARY OUTCOMES:
Scale for Assessment of Negative Symptoms | Baseline, 6M, 12M, 18M, 24M
Scale for Assessment of Positive Symptoms | BL, 6M, 12M, 18M, 24M

CONTACTS AND LOCATIONS:
Overall Officials: Aaron T Beck, MD, Principal Investigator — University Professor, Department of Psychiatry, University of Pennsylvania; Paul M Grant, PhD, Study Director — Assistant Professor, Department of Psychiatry, University of Pennsylvania
Locations (1):
- Psychopathology Resarch Unit, Department of Psychiatry, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Rector NA, Beck AT, Stolar N. The negative symptoms of schizophrenia: a cognitive perspective. Can J Psychiatry. 2005 Apr;50(5):247-57. doi: 10.1177/070674370505000503. PMID 15968839
- [Background] Beck AT, Rector NA, Stolar, NM, & Grant PM. Schizophrenia: Cognitive theory, research, and therapy. New York: Guilford Press
- [Result] Grant PM, Huh GA, Perivoliotis D, Stolar NM, Beck AT. Randomized trial to evaluate the efficacy of cognitive therapy for low-functioning patients with schizophrenia. Arch Gen Psychiatry. 2012 Feb;69(2):121-7. doi: 10.1001/archgenpsychiatry.2011.129. Epub 2011 Oct 3. PMID 21969420
- See also: Beck Institute for Cognitive Therapy and Research — http://www.beckinstitute.org
- See also: National Alliance of Research on Schizophrenia and Depression — http://www.narsad.org/